CLINICAL TRIAL: NCT04077242
Title: Hysteroscopic Evaluation of Fallopian Tubal Patency Compared to Laparoscopic Chromopertubation: a Prospective, Randomized Study on the "Flow" and "Parryscope" Techniques
Brief Title: Hysteroscopic Evaluation of Fallopian Tubal Patency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Johannes Ott, Assoc.Prof. Priv.Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1341/2019
Record Dates: First submitted 2019-08-24; First posted 2019-09-04 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Infertility of Tubal Origin; Infertility, Female; Fallopian Tube Occlusion; Uterus Abnormal
Keywords: hysteroscopy; Parryscope; chromopertubation
MeSH Terms: conditions — Infertility, Female; Uterine Anomalies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Parryscope"-group (Active Comparator): In these patients, Fallopian tube patency is assessed using the "Parryscope" technique. A small amount of air is introduced into the iv tubing by inverting the drip chamber to create air bubbles. When air enters the uterine cavity, a single large air bubble or stream of air bubbles traversing the ostia is considered indicative of tubal patency. At least 10 seconds of intracavitary evaluation is typically performed before air bubble entry to allow pressure equilibration if a hydrosalpinx is present [10]. At least 30 seconds of observation per ostia is performed if patency is not observed.
  Interventions: Diagnostic Test: Hysteroscopic Fallopian tube assessment using the "Parryscope" technique
- "Tubal flow"-group (Active Comparator): In these patients, Fallopian tube patency is assessed using the "flow" technique. a positive "flow" is defined as the observation of saline directly traversing the ostia, endometrial structures floating toward the ostia, or air bubbles traversing the ostia.
  Interventions: Diagnostic Test: Hysteroscopic Fallopian tube assessment using the "Tubal flow" technique

INTERVENTIONS:
Diagnostic Test: Hysteroscopic Fallopian tube assessment using the "Parryscope" technique — A small amount of air is introduced into the iv tubing by inverting the drip chamber to create air bubbles. When air enters the uterine cavity, a single large air bubble or stream of air bubbles traversing the ostia is considered indicative of tubal patency. At least 10 seconds of intracavitary evaluation is typically performed before air bubble entry to allow pressure equilibration if a hydrosalpinx is present [10]. At least 30 seconds of observation per ostia is performed if patency is not observed.
  Arms: "Parryscope"-group
Diagnostic Test: Hysteroscopic Fallopian tube assessment using the "Tubal flow" technique — a positive "flow" is defined as the observation of saline directly traversing the ostia, endometrial structures floating toward the ostia, or air bubbles traversing the ostia.
  Arms: "Tubal flow"-group

SUMMARY:
Hysteroscopy is an important tool in the evaluation of sterility. Assessing tubal patency during hysteroscopy seems highly relevant, particularly when it allows for a low cost, fast, gentle, and accurate way of gathering information that may guide clinical care. Therefore, it is important to know which technique is the best. Thus, the primary aim of this study is to evaluate the reliability of (1.) the hysteroscopic visualization of a "tubal flow" and (2.) the "Parryscope technique" as compared to the gold standard, namely laparoscopic chromopertubation. In a prospective, randomized study, the following women are enrolled: (1.) The patient is subfertile, defined as being unable to become pregnant within a year despite unprotected sexual intercourse. It is also within the standard of care to be presumed subfertile if one has tried for six months and has known risk factors that would hinder conception, including but not limited to anovulation and endometriosis. (2.) A concurrent diagnostic hysteroscopy and laparoscopy with chromopertubation are performed at the Clinical Division of Gynecological Endocrinology and Reproductive Medicine at the Medical University of Vienna. Hysteroscopic evaluation of tubal patency (either by a positive "tubal flow" or a visible flow of air bubbles in the "Parryscope technique") and the result of the laparoscopic chromopertubation (tubal patency existing or not existing) will be the primary outcome parameters. A total 60 patients are enrolled (30 patients in the "flow assessment" group, 30 patients in the "Parryscope" group) and randomization is performed as block randomization in 4 blocks.

DETAILED DESCRIPTION:
Introduction and scientific background:

Hysteroscopy is an important tool in the evaluation of sterility. It allows direct visualization of the uterine cavity and enables the diagnosis of numerous pathologies. Hysteroscopy shows high reliability and is considered the gold standard for intrauterine evaluation.

When performing hysteroscopy, experts often assess the patency of the tubes via the visibility of flow of the hysteroscopic fluid going through the ostia of the tubes. In the recently published study "Assessment of tubal patency: A prospective comparison of diagnostic hysteroscopy and laparoscopic chromopertubation" - it has been demonstrated that visualizing contrasting substances disperse through the ostia is a significant and meaningful metric for tubal patency.

Pre- and posthysteroscopic vaginal sonography for the evaluation of the hysteroscopic fluid in the pouch of Douglas, selective hysteroscopic pertubation of the tubes and the visibility of air bubbles traversing through the Fallopian tube ostia after an air infusion into the uterine cavity have been reported to be reliable methods for hysteroscopic tubal patency assessment. Particularly the last one, also called the "Parryscope technique", named after its inventor, seems to be highly reliable, easy to conduct and clinically relevant. The "Parryscope technique" seems to perform even better than the technique evaluating the "tubal flow".

Assessing tubal patency during hysteroscopy is highly relevant, particularly when it allows for a low cost, fast, gentle, and accurate way of gathering information that may guide clinical care. Therefore, it is important to know which of the above-mentioned techniques is the best. This prospective randomized study aims to compare the hysteroscopic assessment of the tubes via "tubal flow" and the "Parryscope technique".

Study aims:

The primary aim of this study is to evaluate the reliability of (1.) the hysteroscopic visualization of a "tubal flow" and (2.) the "Parryscope technique" as compared to the gold standard, namely laparoscopic chromopertubation.

Study hypotheses:

Null hypothesis: The hysteroscopically visualizable "tubal flow" and the "Parryscope technique" are similarly reliable in the evaluation of tubal patency.

Alternative hypothesis: The hysteroscopically visualizable "tubal flow" shows a lower sensitivity and specificity than the "Parryscope technique" for the evaluation of tubal patency.

Study design:

Prospective, randomized study.

Recruitment:

Women will be invited to participate by medical professionals at the Department of Obstetrics and Gynecology of the Medical University of Vienna using the above mentioned criteria in the course of their admission to the ward one day before surgery. Potential participants are informed about the procedure, clinical relevance and the balance of risk and benefits incurred through study participation. Patients willing to participate will express this through written affirmation (a "consent form").

Additional considerations:

1. Since in the "flow"-group air bubbles might develop spontaneously and, thus, should be assessed, conducting the "Parryscope"-technique is only possible after the evaluation of the tubal flow.
2. Reactive tubal spasms could occur especially during a prolonged hysteroscopy.
3. This is why in one particular patient only one technique should be performed.

Sample size calculation:

The calculation is based upon the following considerations:

1. Direct comparison of the two groups is not possible. Hence, separate evaluation of the two methods will be performed. Evaluating both methods in one particular patient in the course of a single intervention is impossible without a mutual interference (see: "Additional considerations" above).
2. The "flow effect" is considered the less reliable method and thus, the sample size was aligned to this method. An odds ratio of approximately 10, an alpha of 5%, a power of 80%, a general disease likelihood of 39% and a sensitivity of 66% for occluded tubes result in a total amount of 59 tubes and, accordingly, 30 patients.
3. Thus, the group for the "Parryscope"-technique should also contain 59 tubes (= 30 patients).
4. The randomization of the total 60 patients is performed as block randomization in 4 blocks via the software "R".

Statistical analysis:

Numerical data will be reported as mean and standard deviations, nominal variables as number and frequency. The McNemar Test will be used for the calculation of the reliability of the hysteroscopic assessment of the tubes. The sensitivity, specificity, positive and negative predictive values will be provided including the according 95% confidence intervals (95% CI) for both study groups (evaluated technique versus gold standard laparoscopic chromopertubation). Whether the according odds ratio is over 10 will be evaluated by the use of a binary logistic regression model. Statistical analyses were performed with the software "R". Differences were considered significant if p<0.05.

Data quality evaluation:

Extreme values will be double-checked. In addition, a random checks by two independent investigators to ensure the accuracy of the data will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* The patient is subfertile, defined as being unable to become pregnant within a year despite unprotected sexual intercourse. It is also within the standard of care to be presumed subfertile if one has tried for six months and has known risk factors that would hinder conception, including but not limited to anovulation and endometriosis.
* A concurrent diagnostic hysteroscopy and laparoscopy with chromopertubation are performed at the Clinical Division of Gynecological Endocrinology and Reproductive Medicine at the Medical University of Vienna.
* The patient has given her written informed consent after detailed information on the study by medical professionals at the Department of Obstetrics and Gynecology of the Medical University of Vienna.
* The patient is over 18 and under 45 years old.

Exclusion Criteria:

* The patient had a tubectomy on one or both sides.
* There is no "informed consent".
* The patients has active vaginal infection or other conditions that would preclude hysteroscopy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Fallopian tube patency using laparoscopic chromopertubation | In the course of subsequent laparoscopy, i.e. 20-60 minutes after the diagnostic intervention
  tubal patency as assessed by chromopertubation (information provided separately for each side)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Clinical Division of Gynecologic Endocrinology and Reproductive Medicine, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Data will be provided on personal request

REFERENCES:
- [Background] Cholkeri-Singh A, Sasaki KJ. Hysteroscopy for infertile women: a review. J Minim Invasive Gynecol. 2015 Mar-Apr;22(3):353-62. doi: 10.1016/j.jmig.2014.12.163. Epub 2014 Dec 29. PMID 25553895
- [Background] Godinjak Z, Idrizbegovic E. Should diagnostic hysteroscopy be a routine procedure during diagnostic laparoscopy in infertile women? Bosn J Basic Med Sci. 2008 Feb;8(1):44-7. doi: 10.17305/bjbms.2008.2996. PMID 18318671
- [Background] Indraccolo U, Greco P, Scutiero G, Marrocchella S, Sorrentino F, Mastricci L, Matteo M. The role of hysteroscopy in the diagnostic work-up of infertile asymptomatic patients. Clin Exp Obstet Gynecol. 2014;41(2):124-7. PMID 24779234
- [Background] Mahran A, Abdelraheim AR, Eissa A, Gadelrab M. Does laparoscopy still has a role in modern fertility practice? Int J Reprod Biomed. 2017 Dec;15(12):787-794. PMID 29492476
- [Background] Zhang E, Zhang Y, Fang L, Li Q, Gu J. Combined hysterolaparoscopy for the diagnosis of female infertility: a retrospective study of 132 patients in china. Mater Sociomed. 2014 Jun;26(3):156-7. doi: 10.5455/msm.2014.26.156-157. Epub 2014 Jun 21. PMID 25126006
- [Background] Parry JP, Isaacson KB. Hysteroscopy and why macroscopic uterine factors matter for fertility. Fertil Steril. 2019 Aug;112(2):203-210. doi: 10.1016/j.fertnstert.2019.06.031. PMID 31352959
- [Background] Promberger R, Simek IM, Nouri K, Obermaier K, Kurz C, Ott J. Accuracy of Tubal Patency Assessment in Diagnostic Hysteroscopy Compared with Laparoscopy in Infertile Women: A Retrospective Cohort Study. J Minim Invasive Gynecol. 2018 Jul-Aug;25(5):794-799. doi: 10.1016/j.jmig.2017.11.020. Epub 2017 Dec 6. PMID 29221993
- [Background] Hager M, Simek IM, Promberger R, Ott J. The Role of Diagnostic Hysteroscopy in the Evaluation of Fallopian Tube Patency: a Short Review. Geburtshilfe Frauenheilkd. 2019 May;79(5):483-486. doi: 10.1055/a-0826-1326. Epub 2019 May 21. PMID 31148848
- [Background] Habibaj J, Kosova H, Bilali S, Bilali V, Qama D. Comparison between transvaginal sonography after diagnostic hysteroscopy and laparoscopic chromopertubation for the assessment of tubal patency in infertile women. J Clin Ultrasound. 2012 Feb;40(2):68-73. doi: 10.1002/jcu.20883. Epub 2011 Sep 20. PMID 21935964
- [Background] Parry JP, Riche D, Aldred J, Isaacs J, Lutz E, Butler V, Shwayder J. Proximal Tubal Patency Demonstrated Through Air Infusion During Flexible Office Hysteroscopy Is Predictive of Whole Tubal Patency. J Minim Invasive Gynecol. 2017 May-Jun;24(4):646-652. doi: 10.1016/j.jmig.2017.02.010. Epub 2017 Feb 16. PMID 28216455
- [Background] Torok P, Major T. Accuracy of assessment of tubal patency with selective pertubation at office hysteroscopy compared with laparoscopy in infertile women. J Minim Invasive Gynecol. 2012 Sep-Oct;19(5):627-30. doi: 10.1016/j.jmig.2012.03.016. PMID 22935304
- [Background] Parry JP, Riche D, Rushing J, Linton B, Butler V, Lindheim SR. Performing the Parryscope technique gently for office tubal patency assessment. Fertil Steril. 2017 Oct;108(4):718. doi: 10.1016/j.fertnstert.2017.07.1159. Epub 2017 Aug 31. PMID 28843382
- [Background] Hajian-Tilaki K. Sample size estimation in diagnostic test studies of biomedical informatics. J Biomed Inform. 2014 Apr;48:193-204. doi: 10.1016/j.jbi.2014.02.013. Epub 2014 Feb 26. PMID 24582925

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT04077242/Prot_SAP_000.pdf